CLINICAL TRIAL: NCT01771575
Title: The Use of the PoNS™ Device in the Treatment of Blunt and Blast Induced Vestibular Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding received
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: The Geneva Foundation (Other)
Responsible Party: Principal Investigator, Sara Murphy, Research Administrator, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCSD.2013.0011
Record Dates: First submitted 2013-01-14; First posted 2013-01-18 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Hearing and Vestibular Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Experimental): PoNS™ device
  Interventions: Device: PoNS™ device
- Placebo Arm (Placebo Comparator): placebo device
  Interventions: Other: Placebo device

INTERVENTIONS:
Other: Placebo device — Placebo device
  Arms: Placebo Arm
Device: PoNS™ device — The PoNS™ device uses electrotactile waveform in conjunction with the Cranial Nerve - Non-Invasive NeuroModulation (CN-NINM) intervention. This involves using both balance and gait training methods to stabilize symptoms, regain balance & gait, and affect the functional transfer of improved stability and mobility to activities of daily living. It is based on a body of work focused on developing the tongue-based human-machine interface and application of this technology for balance, vision, and auditory substitution and more recently as neuromodulation for brain rehabilitation after injury and disease.
  Other Names: Portable Neuromodulation Stimulator, version 2.2
  Arms: Treatment Arm

SUMMARY:
Traumatic brain injury (TBI) is a major worldwide health issue. Figures from the Centers for Disease control show that 1.7 million people suffer a TBI annually. Meanwhile the World Health Organization recognizes TBI as one of the most significant health issues in developing countries. In the military, mild traumatic brain injury (mTBI) is one of the most frequent sequela of modern war. Dizziness and balance disorders are the most frequent sequela of mTBI and account for a significant degree of mTBI morbidity. At the current time, the best treatment modality for dizziness secondary to mTBI is vestibular rehabilitation (VR). While VR is effective, the therapy is time consuming, not universally successful, and results in incomplete recovery by many patients. Work needs to be done in an attempt to improve therapy outcomes. This project will study the use of neuromodulation (through stimulation of the tongue) as an adjuvant to improve the effectiveness of VR and reduce the time involved in VR. Given past work with variants on this minimal medical impact appliance, using the PoNS™ device to augment therapy may result in a significant improvement in VR outcomes. Given the enormous public health and military burden of mTBI, and given that dizziness is a major component often responsible for significant morbidity, this project has significant military and civilian impact and can be beneficial to those who suffer mTBI worldwide.

DETAILED DESCRIPTION:
The CN-NINM intervention is an experimental regimen. It has been developed over the last 12 years at Tactile Communication and Neurorehabilitation Laboratory (TCNL) at the University of Wisconsin - Madison. All human subjects testing was performed under IRB approval. The PoNS™ is an experimental device that has been evolved over this same period at TCNL, and is not FDA approved. An Investigator's Brochure and attendant Safety Chart have been developed to satisfy requirements for an Investigational Device Exemption, and provide additional context with respect to the research proposed here.

The goal of this work is to test the effectiveness of this device with standard rehabilitation therapy on individuals who have operationally induced balance disorders from blunt or blast head trauma.

SPECIFIC OBJECTIVES:

1. To compare the effectiveness of active PoNS-2 (PoNS™) device combined with standard vestibular rehabilitation to a placebo PoNS™ device with vestibular rehabilitation in patients with blast and blunt head trauma induced dizziness over the time period of a standard course of therapy.
2. To compare the effectiveness of active PoNS™ device combined with standard vestibular rehabilitation to a placebo PoNS™ device with vestibular rehabilitation in patients with blast and blunt head trauma induced dizziness three months after a standard course of rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Head Injury from blunt or blast suffered within the lines of duty
* Not meeting any of the exclusion criteria
* Injury occurred 21 -365 days ago

Exclusion Criteria:

* History of a diagnosed balance disorder prior to injury
* Going through board process before starting participation
* Significant medical issues including but not limited to heart disease, pulmonary disease, autoimmune disorders, severe arthritis, etc.
* Orthopedic injuries that prevent standing and walking
* Age less than 18 or greater than 40 years of age

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Sensory Organization Test score | Change from Baseline SOT score at 3 months
  Posturography for Sensory Organization Test: Utilizing a computerized dynamic posturography (Neurocom Inc., Clackmas, OR) the sensory organization test (SOT) is conducted by measuring postural sway on a force plate under six different conditions as follows 1) Normal Stance eyes open, 2) Normal Stance with eyes closed, 3) Normal Stance with sway referenced visual surround, 4) Sway reference stance eyes open, 5) Sway reference stance with eyes closed, and 6) Sway reference stance with sway referenced vision. The SOT will conduct three trials in each condition and utilize the information to produce a computer generated objective score of balance/posture function. The exam takes less than ten minutes to produce.

SECONDARY OUTCOMES:
Change in Vestibular-Ocular Reflex scores | Change from Baseline VOR score at 3 months
  VOR Tests: A Neuro Kinetics IPortal Video-oculography system (Neurokinetics Inc., Pittsburgh, PA) with a six degree of freedom accelerometer will be used to (1) document head thrust test findings qualitatively and (2) provide objective measurements of test results. The software will be configured for (1) detection of head thrusts of appropriate direction and orientation (re: earth vertical) and (2) real-time determination of performance parameters (VOR).

OTHER OUTCOMES:
Change in Functional Gait Assessment Test scores | Change from Baseline FGAT score at 3 months
  The Functional Gait Assessment Test (FGAT) is a 10 item gait task test in which each task is graded on a 0-3 scale with 0 indicating could not perform and 3 indicating performed without error. Grading is done by an experienced rater. The FGAT produces an ordinal score on a 0-30 point scale and is normed from previous civilian and military studies.
Change in Dizziness Handicap Index scores | Change from Baseline DHI score at 3 months
  The Dizziness Handicap Index (DHI) is a well-validated self report the produces a score on a hundred-point scale.
Change in Activities specific Balance Confidence scale scores | Change from Baseline ABC score at 3 months
  The Activities specific Balance Confidence scale (ABC) is a 16 question survey in which individuals' answer how confident they are about being able to perform a balance related task on a 0%-100% scale. The questionnaire is scored by adding the percentages and dividing by 100% to arrive at a scaled score form 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Hoffer, M.D., Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No